CLINICAL TRIAL: NCT06022601
Title: Post Delivery Intervention in Women With Previous Gestational Diabetes Mellitus to Improve Glycaemia
Acronym: Post-GDM-DNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 292085
Record Dates: First submitted 2023-06-06; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNA Nudge (Experimental): DNA Nudge wearable and app, DNA-based dietary advice
  Interventions: Device: DNA Nudge
- Control (No Intervention): Fitbit, standard dietary advice

INTERVENTIONS:
Device: DNA Nudge — DNA Nudge wearable, DNA-based dietary advice
  Arms: DNA Nudge

SUMMARY:
STUDY SUMMARY

TITLE Post-delivery intervention in women with previous gestational diabetes mellitus for weight loss, glycaemia and cardiovascular health DESIGN Feasibility study Allocation: RCT AIMS To determine the feasibility of a post-delivery intervention to improve glycemia and cardiovascular function and promote weight loss in women who have had gestational diabetes.

OUTCOME MEASURES Primary outcome; Effect of intervention on HbA1c: difference in HbA1c between intervention arm and control arm measured at 12 weeks.

Secondary Outcomes;

* Adherence to intervention;
* Willingness to be randomised to post-delivery intervention;
* Process measures to evaluate patient experience of study and intervention;
* Participants' preferred time to commence the study, within the start date allowance of 6 weeks - 6 month post-delivery.
* Between-arm differences and within-arm differences to evaluate:

  * Effect of intervention on HbA1c at 12 and 24 weeks
  * Effect of intervention on weight and BMI at 12 and 24 weeks
  * Effect of intervention on systolic and diastolic blood pressure at 12 and 24 weeks
  * Effect of intervention on lipid profile (total cholesterol, HDL, LDL) at 12 and 24 weeks
  * Effect of intervention on physical activity at 12 and 24 weeks POPULATION We will recruit 50 women aged 18-45 with previous gestational diabetes and randomise them to 1 of 2 arms to commence study at 6 weeks - 6 months post-delivery. Women starting the study at 13 weeks post-delivery will have their routine post-delivery HbA1c act as baseline HBA1c.

ELIGIBILITY Pregnant women with gestational diabetes (women will be given the option to start the study between 6 weeks and 6 months post-delivery) or women who have given birth in the last 12 months and had gestational diabetes during that pregnancy; aged 18-45; and access to a smartphone with an operating system of iOS 9.0 or above, or Android 5.0 or above.

DURATION Study duration: 1/4/21-1/9/22. Participant duration: 24 weeks

DETAILED DESCRIPTION:
STUDY OBJECTIVES Objectives

To assess:

1. Effect of intervention on HbA1c at 12 and 24 weeks
2. Adherence to intervention
3. Participants' preferred time to commence the study, within the start date allowance of 6 weeks - 6 month post-delivery.
4. Qualitative data on how participants found post-delivery intervention
5. Effect of intervention on weight at 12 and 24 weeks
6. Effect of intervention on systolic and diastolic blood pressure at 12 and 24 weeks
7. Effect of intervention on lipid profile (total cholesterol, HDL, LDL) at 12 and 24 weeks
8. Effect of intervention on physical activity at 12 and 24 weeks

3. STUDY DESIGN We will conduct a feasibility study for an open-label, randomised, controlled trial of a personalised post-delivery intervention (DNA Nudge) to improve weight, glycaemia and cardiovascular function in women with previous GDM.

The study is designed to be remote, to enable the study to begin and continue in the pandemic and minimise barriers to recruitment. Study participants will be provided with equipment and instructions to collect samples and measurements at home. Contact with the research team will be over telephone or Microsoft Teams video call.

We will advertise in diabetes antenatal clinics using word-of-mouth, posters, social media and on departmental emails at Imperial College Healthcare NHS Trust or Imperial College for women with current/previous GDM aged 18-45. We will recruit via Twitter, email and in-person encounters.

We will randomise women to 1 of 2 arms:

Arm 1: Standard dietary and physical activity advice as per NICE guidelines at week 1 (active control arm; n = 25) Arm 2: DNA-based personalised dietary and physical advice delivered by DNA Nudge dietician at week 1 and by DNA Nudge wearable and app for weeks 1-24 (intervention arm; n = 25)

Women not randomised to DNA Nudge will be provided with an activity app/wearable device (Fitbit) to monitor daily step count. All women will be provided with a home BP monitor and weighing scales.

Week 1 Eligibility assessment, consent, randomisation, IPAQ questionnaire, baseline BP and weight, blood sample collected for baseline lipid profile.

Some women will begin the study at 13 weeks post-delivery and coincide with the routine postnatal HbA1c for women with GDM. The routine post-delivery HbA1c will be baseline HbA1c for this study. For women who commence the study outside the 13 weeks post-delivery window, a finger prick blood sample will be used for a baseline HbA1c test.

Women in the control arm will be given standard dietary and physical activity advice by the research team, in line with NICE guidelines.

Women in the DNA Nudge arm will provide a cheek swab for DNA analysis, carried out by DNA Nudge. They will be given personalised dietary advice by a DNA Nudge dietician, and be provided with DNA Nudge wearable, app and instructions.

Week 6:

Telephone/video-call follow-up to check ongoing willingness to participate and assess adherence.

Week 12:

Collect weight and BP data from weeks 1-12, collect blood sample for HbA1c and lipid profile. Check ongoing willingness to participate and assess adherence.

Week 18:

Telephone/video-call follow-up to check ongoing willingness to participate and assess adherence.

Week 24:

Collect weight and BP data from weeks 12-24, follow-up IPAQ questionnaire, collect blood sample for HbA1c and lipid profile, return devices and collect usage data from DNA Nudge. Qualitative questionnaire to explore intervention experience.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational diabetes (women will be given the option to start the study between 6 weeks and 6 months post-delivery) or
* women who have given birth in the last 12 months and had gestational diabetes during that pregnancy
* aged 18-45,
* access to a smartphone with an operating system of iOS 9.0 or above, or Android 5.0 or above

Exclusion Criteria:

* Diabetes outside of pregnancy (diagnosis of type 1 or 2 diabetes; or HbA1c 48 mmol/mol or above).
* Health contra-indications to moderate-vigorous exercise.
* Planning pregnancy during the study period or become pregnant during the study period. -Cancer
* kidney disease
* liver disease
* pancreatitis.
* gastric bypass surgery or similar weight loss surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Glycaemia

SECONDARY OUTCOMES:
HbA1c | 24 weeks
  Glycaemia
Weight | 12 weeks
  kg
Weight | 24 weeks
  kg
Systolic and diastolic Blood pressure | 12 weeks
  mmHg
Systolic and Diastolic Blood pressure | 24 weeks
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request from the PI
Supporting Information: Study Protocol, ICF

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06022601/Prot_SAP_000.pdf